CLINICAL TRIAL: NCT06540976
Title: Posterior Cingulate Cortex and Executive Control of Episodic Memory
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R01MH129439 (NIH)
Record Dates: First submitted 2024-04-16; First posted 2024-08-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Episodic Memory
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experiment 1 - episodic / executive switch (Experimental): All enrolled participants will be asked to perform experiment 1, which is a cognitive task involving the switch between performing episodic memory decisions (e.g., "did you eat fruit yesterday?") and executive decisions (e.g. "...does 5+3+8 = 17?"). Participants will perform this computer-based task while electrical brain activity is recorded from the posterior cingulate cortex, hippocampus and prefrontal cortex. This task takes 18 minutes to complete.
  Interventions: Behavioral: Cognitive testing
- Experiment 2 - executive decision task (Experimental): All enrolled participants will be asked to perform experiment 2, which is a cognitive task involving reward-based decisions between two options. For each decision, the two options will differ in their risk and reward (e.g., 100% chance of 10 points vs. 30% chance of 50 points). Participants will perform this computer-based task while electrical brain activity is recorded from the posterior cingulate cortex, hippocampus and prefrontal cortex. This task takes 15 minutes to complete.
  Interventions: Behavioral: Cognitive testing
- Experiment 3 - episodic decision task (Experimental): All enrolled participants will be asked to perform experiment 3, which is a cognitive task involving memory-based decisions between two options (pictures of people). For each decision, the two pictures will differ in memory strength and reward (e.g., familiar picture for 10 points vs. unfamiliar picture 50 points). Memory strength for each picture will be defined by how many times the picture was previously shown (e.g., 2 vs. 10 presentations) prior to performing the memory decision task. Participants will perform this computer-based task while electrical brain activity is recorded from the posterior cingulate cortex, hippocampus and prefrontal cortex. This task takes 15 minutes to complete.
  Interventions: Behavioral: Cognitive testing

INTERVENTIONS:
Behavioral: Cognitive testing — Cognitive tasks testing executive and episodic based decisions, and the switching between these processes.

SUMMARY:
This project will use intracranial recordings and stimulation of the human brain to understand the unique contributions of the posterior cingulate cortex (PCC) to episodic memory behavior. The goal is to test how distinct subregions of the PCC differentially contribute to memory-based decisions (e.g., have I seen this picture before?). The ability to perform invasive studies of the human brain is through routine clinical monitoring of brain activity which occurs during the neurosurgical treatment of epilepsy. However, this project only focuses on the basic science of PCC and memory behavior. Specifically, the investigators will use single-0cell and population measures of brain activity to test a new theory of PCC function which focuses on the executive processes needed to support memory retrieval and memory-based decisions. By studying the PCC, a convergence zone of memory and executive brain systems, progress can be made in elucidating how the failure to successfully leverage past experiences in daily behavior can occur as a common symptom of both neurodegenerative disease (e.g., Alzheimer's disease) and multiple psychiatric conditions (e.g., schizophrenia) implicating PCC dysfunction.

DETAILED DESCRIPTION:
This project reflects a basic experimental study involving human participants (BESH), which focuses on the neuroscience of episodic memory. Episodic memory involves the encoding and retrieval of past experiences to support learned behavior. Aside from these mnemonic processes, it also requires the ability to regulate memory (i.e. executive processes). For example, many real-world decisions will engage episodic retrieval, for which executive processes must help to integrate and evaluate the quality of remembered information (mnemonic evidence) and guide behavior to either decision, action, or continued memory search. While the neural basis of episodic memory encoding and retrieval have been a major focus of research, far less is known about its executive aspects. Executive mnemonic functions likely involve an anatomical substrate that is (i) multisensory/associative, (ii) engaged by memory/executive processing, and (iii) strongly interconnected with both mnemonic regions in the medial temporal lobe (MTL) and executive prefrontal (PFC) regions. Prior non-human primate studies, as well as human electrophysiology and neuroimaging data, suggest that posterior cingulate cortex (PCC) fulfills these criteria. The central hypothesis of this work is that the PCC plays a critical and unique role in executive control of episodic memory retrieval. The investigators further hypothesize that it comprises three subregions regions: dorsal PCC, ventral PCC and retrosplenial cortex (RSC). These subregions are proposed to play complementary roles, corresponding to retrieval regulation, retrieval integration, and scene perception and transformation, respectively. In this account, PCC is a convergence zone of memory and executive systems, whose specific functional organization accounts for prior discrepancies between studies and species. The investigators will utilize human intracranial recordings, including single-cell data and stimulation within PCC, to better resolve the functional organization of this region. The investigators will employ an array of cognitive experiments to delineate three PCC subregions supporting the encoding, retrieval and executive control of memory processing (Aim 1). In delineating these subregions, the investigators will also seek to differentiate PCC responses from those occurring in memory and executive functional networks (Aim 2). Finally, based on these observations, the investigators will demonstrate the causal role of PCC subregions on behavior and local/network activity (Aim 3). By studying PCC, a convergence zone of memory and executive systems, progress can be made in elucidating how the failure to successfully leverage past experiences in daily behavior can occur as a common symptom of both neurodegenerative disease (e.g. Alzheimer's disease) and multiple psychiatric conditions (e.g. schizophrenia) implicating PCC dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* All participants are patients undergoing invasive brain monitoring for epilepsy and will be asked to consent to participation in this basic science protocol (which is focused on the patient group but is not focused on the study of epilepsy).

Exclusion Criteria:

* Individuals not undergoing invasive brain monitoring for epilepsy.
* Individuals outside of the age range (18-50 yrs).
* Individuals with cognitive impairment or intellectual difficulty.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2027-03-02 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Episodic/Executive behavioral task performance accuracy | Outcome assessed 10 minutes after intervention
  Participants will perform three tasks each testing the accuracy of executive (reward) or episodic (memory strength) based decisions. Outcome measures will be decision accuracy (% correct).
Episodic/Executive behavioral task performance speed | Outcome assessed 10 minutes after intervention
  Participants will perform three tasks each testing the speed of executive (reward) or episodic (memory strength) based decisions. Outcome measures will be response/decision reaction time (milliseconds).
Changes in high-frequency electrophysiological brain response | Outcome assessed 1 hour after intervention
  During behavioral task performance, electrophysiological signals recorded from the brain will be quantified for changes in the mean high-frequency activity (70-150 Hz) amplitude during correct and incorrect episodic/executive decisions. The goal is to track this electrophysiological activity to quantify if and when brain activity in the posterior cingulate cortex occurs during memory and non-memory based decisions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania - Pavilion, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the National Institute of Mental Health Data Archive (NIMH NDA).
Supporting Information: Analytic Code